CLINICAL TRIAL: NCT05197361
Title: Evolución de Las Resistencias Microvasculares y Del Flujo Coronario Absoluto en Pacientes Con intervención Coronaria percutánea de Una oclusión crónica
Brief Title: Microvascular Coronary Resistance and Absolute Coronary FLOW in Patients With Percutaneous Intervention of a Chronic Total Occlusion
Acronym: FLOW-CTO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Other Study IDs: FLOW1
Record Dates: First submitted 2022-01-05; First posted 2022-01-19 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Chronic Total Occlusion of Coronary Artery; Microvascular Coronary Artery Disease; Coronary; Ischemic; Coronary Microvascular Dysfunction
MeSH Terms: conditions — Ischemia | interventions — Fractional Flow Reserve, Myocardial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Global cohort: Invasive coronary physiology parameters estimation, including:
  FFR, CFR, IMR, Absolute coronary flow (AF). AF derived resistances
  Interventions: Diagnostic Test: Invasive coronary physiology

INTERVENTIONS:
Diagnostic Test: Invasive coronary physiology — Estimation of guide-wire coronary physiology parameters
  Other Names: fractional flow reserve; coronary flow reserve; index of microvascular resistance; absolute coronary flow; AF-derived coronary resistance

SUMMARY:
It is an observational study which objective is to analyze, through a series of invasive parameters, the state of the coronary microvasculature immediately after the successful percutaneous coronary intervention of a chronic total occlusion and at 6 months after the index procedure.

The aim of the study is to check the variation in the values of the index of microcirculatory resistance (IMR) and invasive absolute coronary flow (AF). The working hypothesis is that, in the follow-up of these patients, AF will increase significantly with respect to its baseline and, conversely, IMR will be reduced during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Those patients with a clinical indication for percutaneous coronary intervention of a chronic total occlusion. As a routine clinical practice in our center, it is proposed to perform a angiographic follow-up 6 months after the index procedure.

Exclusion Criteria:

* No specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic heart disease and evidence of at least one chronic total occlusion, with data of inducible ischemia and/or viability and susceptible to percutaneous coronary intervention.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Variation in the values of IMR between basal and 6-months follow-up | 6 months
Variation in the values of absolute coronary flow between basal and 6-months follow-up | 6 months

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital del Mar, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Puerta del Mar, Cadiz
  - Hospital Universitario de La Princesa, Madrid

IPD SHARING:
Plan to Share IPD: Undecided